CLINICAL TRIAL: NCT07289373
Title: Moderate Intensity Training Versus High Intensity Interval Training on Gait and Energy Expenditure in Children With Spastic Diplegia.
Brief Title: Moderate Versus High-intensity Interval Training in Children With Diplegia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Assisstant Proffessor, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002427
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A (received aerobic training with moderate intensity endurance training "MIET" by walking or running on a treadmill). Treatment was delivered for 20minutes, 3 times per week for two successive months.
  Interventions: Procedure: Moderate intensity training
- Group B (Experimental): Group B (received aerobic training exercises in the form of high-intensity interval training (HIT) by walking or running on a treadmill). Treatment was delivered for 20minutes, 3 times per week for two successive months.
  Interventions: Procedure: High intensity interval training

INTERVENTIONS:
Procedure: Moderate intensity training — Moderate-intensity endurance training (MIET) by walking or running on a treadmill
  Arms: Group A
Procedure: High intensity interval training — Aerobic training exercises in a form of high-intensity interval training (HIIT) by walking or running on a treadmill
  Arms: Group B

SUMMARY:
The aim is to compare the effects of moderate-intensity training and high-intensity interval training on gait, energy expenditure, and functional mobility in children with spastic diplegia. Methods: Thirty children with spastic diplegic cerebral palsy were allocated randomly into two groups (n=15 each). The group A and the group B. Assessment of functional mobility and energy expenditure and gait analysis for all children of both groups were assessed before and after the suggested period of treatment.

DETAILED DESCRIPTION:
Methods: Thirty children with with spastic diplegic cerebral palsy were allocated randomly into two groups ( n= 15 each). The group A (received aerobic training with moderate intensity endurance training "MIET" by walking or running on a treadmill) and the group B (received aerobic training exercises in a form of high intensity interval training "HIT" by walking or running on a treadmill). Treatment was delivered for 20minutes, 3 times per week for two successive months. Assessment of functional mobility and energy expenditure using Timed Up and Go(TUG) test and Energy Expenditure Index Heart Rate(EEIHR) respectively, while gait analysis for both lower limb angles of (hips and Knees) assessment using 2d gait analysis by( Kinovea) software. All children of both groups assessed before and after the suggested period of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Their age ranged from 3 to 5 years old
2. The degree of spasticity ranged from 1+ to 2 according to modified Ashworth scale
3. They were able to walk with limitations or holding on according to Gross Motor Function Classification System (II, III).
4. They were able to follow instructions and understand commands.
5. They were medically stable.

Exclusion criteria:

1. Children who had bone and tendon lengthening surgeries within the last 6 months.
2. Children with lung and heart diseases and disorders.
3. Children with fixed deformities in joints and bones of lower limbs.
4. Children performing different sorts of physical activities.
5. Children receiving any medications affecting muscle and mental function or antiepileptic drugs that affect the mental function.
6. Children with perceptual defects.
7. Children with any visual or sound-related issues.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Gait | 2 months
  Assessed by 2D gait analysis
Functional mobility | 2 months
  Assessed by Time Up and Go test
Energy Expenditure | 2 months
  Assessed by Energy Expenditure Index Heart Rate

CONTACTS AND LOCATIONS:
Overall Officials: Mai E. Abbass, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No